CLINICAL TRIAL: NCT01220167
Title: Open-label, Randomized, Three-way Crossover Bioavailability Study Comparing Ondansetron Orally Dissolving Filmstrip (ODFS) With and Without Water to Zofran Orally Dissolving Tablets (ODT) Without Water in Healthy Adult Study Participants
Brief Title: Three-way Crossover Study Comparing Ondansetron ODFS Administered With and Without Water to Zofran ODT Without Water
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aquestive Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OND/CR/051/08/09
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Healthy Participants
Keywords: bioavailability
MeSH Terms: interventions — Ondansetron; Water

STUDY DESIGN:
Intervention Model Description: Open label, balanced, randomized three period, three treatment, three sequence, three-way crossover bioavailability study .
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence ABC (Experimental): Six subjects received a single dose of each of the 3 study treatments in the following order: Test Treatment A (Ondansetron 8 mg ODFS without water), Test Treatment B (Ondansetron 8 mg ODFS with water), Test Treatment C (Zofran ODT® containing ondansetron 8 mg without water). Each dose was administered following a 10-hour fast with a 3-day washout period between doses.
  Interventions: Drug: Ondansetron 8 mg ODFS without water; Drug: Ondansetron 8 mg ODFS with water; Drug: Zofran ODT (ondansetron 8 mg) without water
- Sequence BCA (Experimental): Six subjects received a single dose of each of the 3 study treatments in the following order: Test Treatment B (Ondansetron 8 mg ODFS with water), Test Treatment C (Zofran ODT® containing ondansetron 8 mg without water), Test Treatment A (Ondansetron 8 mg ODFS without water). Each dose was administered following a 10-hour fast with a 3-day washout period between doses.
  Interventions: Drug: Ondansetron 8 mg ODFS without water; Drug: Ondansetron 8 mg ODFS with water; Drug: Zofran ODT (ondansetron 8 mg) without water
- Sequence CAB (Experimental): Six subjects received a single dose of each of the 3 study treatments in the following order: Test Treatment C (Zofran ODT® containing ondansetron 8 mg without water), Test Treatment A (Ondansetron 8 mg ODFS without water), Test Treatment B (Ondansetron 8 mg ODFS with water). Each dose was administered following a 10-hour fast with a 3-day washout period between doses.
  Interventions: Drug: Ondansetron 8 mg ODFS without water; Drug: Ondansetron 8 mg ODFS with water; Drug: Zofran ODT (ondansetron 8 mg) without water

INTERVENTIONS:
Drug: Ondansetron 8 mg ODFS without water — Single dose of Ondansetron 8 mg (ODFS) administered without water
  Other Names: Test Treatment (A)
Drug: Ondansetron 8 mg ODFS with water — Single dose of Ondansetron 8 mg (ODSF) was orally administered, allowed to dissolve, swallowed with saliva, followed with water
  Other Names: Test Treatment (B)
Drug: Zofran ODT (ondansetron 8 mg) without water — Single dose of Zofran ODT (containing ondansetron 8 mg) administered without water
  Other Names: Reference Treatment (C)

SUMMARY:
This study conducted in healthy male and female adult participants compared the bioavailability and relative safety and tolerance of a single dose of ondansetron 8 mg Orally Dissolving Filmstrip (ODFS) administered under fasting conditions with and without water with that of a single dose of Zofran Orally Dissolving Tablets (ODT®) containing ondansetron 8 mg administered under fasting conditions without water.

DETAILED DESCRIPTION:
This was an open-label, single oral dose,randomized sequence, three-way crossover study to compare the bioavailability, safety and tolerability of ondansetron 8 mg Orally Dissolving Filmstrip (ODFS) administered without (Test Treatment A) and with water (Test Treatment B) with that of Zofran Orally Dissolving Tablets (ODT®) containing ondansetron 8 mg administered without water (Reference Treatment C) in healthy adult participants. The 3 treatment sequences were: ABC, BCA, and CAB, in which, all treatments were administered after an overnight fasting of at least 10 hours in each period.

Participants reported to the study site between 07:30 am to 04:30 pm on 22 Aug 2008, 25 Aug 2008, and 28 Aug 2008 for Period 1, Period 2, & Period 3, respectively. Participants were served dinner between 8:00 pm to 8:30 pm, to ensure a minimum of 10 hours of fasting prior to administration of a single dose of either the test or reference product. Participants were dosed as per the randomization schedule with a 3-day wash out period between each administration.

A total of 18 blood samples (4 mL each) were collected from each subject in each period for pharmacokinetic analyses. Safety assessments including monitoring of adverse events, periodic physical examination, and vital signs monitoring. Urine Drug Screening was done at the time of check-in of all the study periods to identify participants with any substance abuse. Urine pregnancy screen (for female subjects only) was scheduled at the time of screening and at admission for Period 1, Period 2, Period 3. A clinical assessment, which included general and systemic examination, was done at the pre-study screening and post study physical examination. Clinical laboratory hematology and chemistry tests were performed at screening (pre-study) and at the study follow-up visit (post-study).

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion in the study were:

* Study volunteer should provide written informed consent.
* Study volunteer must be a healthy adult within 18-45 years of age (inclusive).
* Study volunteer should have a Body mass index of ≥ 18.5 kg/m2 and ≤ 25 kg/m2, with body weight not less than 50 kg.
* Study volunteer should have a systolic blood pressure with upper limit of less than 140 mmHg and lower limit of more than or equal to 90 mm Hg.
* Study volunteer must be of normal health as determined by medical history and physical examination performed within 15 days prior to the dosing of period 1.
* Study volunteer should have a normal ECG, chest X-ray and vital signs.
* If study volunteer is a female and is of child bearing potential she must be practicing an acceptable method of birth control for the duration of the study.

Exclusion Criteria:

The criteria for exclusion from the study were:

* Study volunteer incapable of understanding the informed consent.
* Study volunteer with a history of hypersensitivity or idiosyncratic reaction to study drug or any other related drug.
* Study volunteer having any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
* Study volunteers with a history of tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma
* Study volunteer who smokes regularly more than ten cigarettes daily.
* Study volunteer who has taken over the counter or prescribed medications.
* Study volunteer with a history of any psychiatric illness, which may impair the ability to provide written, informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudershan Vishwanath, MD, Principal Investigator — Vimta Labs Ltd.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-five healthy adult volunteers were screened for study eligibility between 18 Aug 2008 and 21 Aug 2008 at VIMTA VHS Research Centre in Adyar, Chennai - 600 113, India.
Pre-assignment Details: Eighteen of 55 subjects were randomized. Of those not randomized, 29 did not meet eligibility criteria and 6 declined to participate. The 18 eligible participants reported to the study site on 22 Aug 2008, 25 Aug 2008 and 28 Aug 2008 for Period 1, Period 2, & Period 3, respectively.
Groups:
- Sequence ABC: Each subject received a single dose of each of the 3 study treatments in the following order: Test Treatment A (Ondansetron 8 mg ODFS without water), Test Treatment B (Ondansetron 8 mg ODFS with water), Test Treatment C (Zofran ODT containing ondansetron 8 mg without water).
- Sequence BCA: Each subject received a single dose of each of the 3 study treatments in the following order: Test Treatment B (Ondansetron 8 mg ODFS with water), Test Treatment C (Zofran ODT containing ondansetron 8 mg without water), Test Treatment A (Ondansetron 8 mg ODFS without water).
- Sequence CAB: Each subject received a single dose of each of the 3 study treatments in the following order: Test Treatment C (Zofran ODT containing ondansetron 8 mg without water), Test Treatment A (Ondansetron 8 mg ODFS without water), Test Treatment B (Ondansetron 8 mg ODFS with water).
Period: Period 1
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB
Started | 6 | 6 | 6
Completed | 6 | 5 | 6
Not Completed | 0 | 1 | 0
Not completed — Urine positive for substance abuse | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 27.6 (7.57) | 31.1 (8.27) | 28.8 (5.98) | 28.2 (6.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 4 | 4 | 6 | 14
Body Mass Index (kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (0.07) | 22.8 (0.78) | 22.9 (1.95) | 23.7 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum Plasma Concentration (Time to reach maximum concentration)
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: 18 subjects were enrolled. One subject did not complete.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ondansetron ODFS With or Without Water and Zofran ODT: Single dose of Ondansetron ODFS 8 mg film administered with and then without water and Zofran 8 mg administered without water
Arm/Group | Ondansetron ODFS With or Without Water and Zofran ODT
Number analyzed (Participants) | 18
ng/mL
  ODFS without water: number analyzed (Participants) | 17
  ODFS without water | 40.866 (13.3089)
  ODFS with water | 42.843 (15.9103)
  Zofran ODT | 39.382 (12.3572)

2. Primary Outcome: AUCt
Description: Area Under Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (e.g., "0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose")
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: 18 healthy subjects were enrolled. Only 17 subjects completed the study. 0 to 96 hours post-dose
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Ondansetron ODFS With and Without Water and Zofran ODT: Single dose of Ondansetron ODFS 8 mg film with and again without water and Zofran 8 mg without water
Arm/Group | Ondansetron ODFS With and Without Water and Zofran ODT
Number analyzed (Participants) | 17
ng*hr/mL
  ODFS without water | 290.687 (106.5203)
  ODFS with water | 291.069 (99.5911)
  Zofran ODT | 285.457 (105.3048)

3. Primary Outcome: AUCinf
Description: Area Under Plasma Concentration-Time Curve From Time Zero to Time Infinity
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: 18 subject were enrolled. Only 17 completed the study.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Ondansetron ODFS With and Without Water and Zofran ODT: Single dose of Ondansetron ODFS 8 mg film with water and without water and Zofran 8 mg without water
Arm/Group | Ondansetron ODFS With and Without Water and Zofran ODT
Number analyzed (Participants) | 17
ng*hr/mL
  ODFS without water | 311.349 (119.7910)
  ODFS with water | 310.394 (112.7499)
  Zofran ODT | 306.497 (121.8256)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of the first dose until 30 days following the last dose (overall approximately 1.5 months for each subject). No adverse events were reported during the study and follow-up period. Clinical laboratory hematology and chemistry tests were performed at screening (pre-study) and at the study follow-up visit (post-study). Thus, abnormal laboratory analytes reported as adverse events could not be attributed to any of the 3 study treatments.
Description: All adverse events (AE) were recorded from the time of the first dose until the last follow-up visit scheduled 48 hours following the last dose of study intervention. Serious adverse events (SAEs) were reported from the time of the first dose until 30 days following the last dose.
  Subjects with AEs considered related to study drug and any SAE regardless of causality were followed until resolution of the event or the subject was lost to follow-up.
Groups:
- ODFS 8 mg With and Without Water and Zofran ODT Without Water: Single dose of ondansetron ODFS 8 mg film administered with and without water and Zofran 8 mg administered without water in randomized sequence.
  Clinical laboratory hematology and chemistry tests were performed at screening (pre-study) and at the study follow-up visit (post-study). Thus, abnormal laboratory analytes reported as adverse events could not be attributed to any of the 3 study treatments.
Arm/Group | ODFS 8 mg With and Without Water and Zofran ODT Without Water
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ODFS 8 mg With and Without Water and Zofran ODT Without Water (N=18)
Alanine aminotransferase increase (Hepatobiliary disorders) | 3 (3) — ALT increased
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1) — AST increased
White blood count increased (Investigations) | 1 (1) — WBC count increased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes